CLINICAL TRIAL: NCT02704546
Title: The Effect of the Drug Methylphenidate on Physiological Stress and Function During Exposure to Exercise and Heat Stress in ADD/ADHD Treated Patients
Brief Title: Methylphenidate (Ritalin®) Effect During Exposure to Exercise and Heat Stress in ADD/ADHD Treated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SHEBA-14-1245-HS-CTIL
Record Dates: First submitted 2016-03-06; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Methylphenidate
MeSH Terms: interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Experimental): In experimental days taking MPH, subjects will take 20mg Ritalin® (Novartis AG) in two tablets of 10mg, by swallow 1 hour prior to performing the physical test.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): In experimental days with placebo subjects will be asked to ingest 2 capsules identical to Ritalin® capsules, by swallow 1 hour prior to performing the physical test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — oral capsules (per os) each containing 10mg Methylphenidate.
  Other Names: Ritalin®, MPH
  Arms: Methylphenidate
Drug: Placebo — capsules identical in shape, colour and size to the Ritalin® capsules, which contain only the inactive ingredients of the same formulation.
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the possible effects of MPH use on physiological functions among ADHD\ADD patients, by performing a set of physical trials to assess aerobic and anaerobic capacity, to characterize the tendency for muscle break down while performing monitored moderate physical effort and to assess the physiological strain while performing moderate exercise in heat load conditions by using the heat tolerance test.

DETAILED DESCRIPTION:
20 male, non-combat soldiers with a pre-existing childhood diagnosis of ADHD\ADD, who are chronically treated with MPH will participate in the study. If necessary, civilian volunteers with a childhood diagnosis of ADHD\ADD may also be recruited to complete the study population (up to 50%, i.e. 10 participants).

1. st encounter: the subjects will receive an explanation of the study and sign an informed consent form, complete a medical questionnaire and undergo physical examination by a physician, including ECG.
2. nd-9th encounter: the subjects will be requested to undergo 10 tests on 8 examination days, which will include the: maximal oxygen consumption test, wingate test, heat tolerance test and step test. Each subject will perform each test twice: once while taking MPH and once with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Civilian volunteers aged 18-25 years.
* BMI range of 17-25.
* Diagnosed with attention deficit disorder (ADD or ADHD) since childhood.
* Routine use of Methylphenidate (at least 5 days a week).
* Without known medical illness or medication use.
* Report of performing physical exercise (twice or more a week).
* Without history of heat injury.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Infectious disease 3 days prior to the experiment.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
physiological strain (composite) | 2 experimental days for each participant
  the physiological strain will be determined by monitoring body core temperature and heart rate of the subjects during a Heat Tolerant Test (HTT). the test is performed in a climatic chamber. during the test the subjects walks on a treadmill (5 km/h and 2% incline) for 2h.
aerobic capacity | 2 experimental days for each participant
  the aerobic capacity of the subjects will be determined by performing a maximal oxygen consumption test (VO2max). VO2 will be monitored continuously with a metabolic system (ERGOTEST 680, ZAN, GERMANY ).

SECONDARY OUTCOMES:
Rectal temperature | 2 experimental days for each participant
  rectal temperature will be recorded at a depth of 10 mm past the anal sphincter using YSI-401 thermal thermistor during each heat tolerance test (HTT).
skin temperature | 2 experimental days for each participant
  The skin temperature will be monitored by skin thermistors located at 3 sites (chest, arm and leg).
heart rate | 8 experimental days for each participant
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
lactic acid | 8 experimental days for each participant
  lactic acid level is assessed from blood drop (finger sting), will be taken before and after every test. lactic acid is a marker for anaerobic effort evaluating.

CONTACTS AND LOCATIONS:
Overall Officials: Haggai Schermann, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel

IPD SHARING:
Plan to Share IPD: No